CLINICAL TRIAL: NCT07022145
Title: A Real-World Multicenter, Prospective, Non-Randomized Parallel Controlled Study on the Optimal Endovascular Therapy for Improving Distal Perfusion and Remodeling of Acute Type B Aortic Dissection
Brief Title: Real-World Prospective Parallel Controlled Study on Endovascular Therapy for Improving Perfusion and Remodeling of TBAD
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Zhihui Dong, Professor, Shanghai Zhongshan Hospital
Other Study IDs: 2023ZD-TEVAR-DBS
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Type B Aortic Dissection
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PSG: Type B aortic dissection patients treated with proximal stent-graft
  Interventions: Procedure: Endovascular repair
- PSG+DBS: Type B aortic dissection patients treated with proximal stent-graft combined with distal bare stent
  Interventions: Procedure: Endovascular repair

INTERVENTIONS:
Procedure: Endovascular repair — Endovascular repair using proximal stent-graft or proximal stent-graft combined with distal stent for TBAD patients

SUMMARY:
There are both common and individual characteristics in patients with type B aortic dissection. Currently, for all subtypes of acute type B dissection, proximal endovascular repair is mostly performed during the subacute phase, while the distal dissection of the descending aorta is often managed with a "watch and wait" strategy. However, such a uniform approach carries potential risks, including imprecise indications, inappropriate timing, and uncertain prognosis. Our research team has previously established a comprehensive database and imaging repository of nearly 10,000 cases of type B dissection. Building upon existing subtypes-such as acute complicated, uncomplicated, penetrating atherosclerotic ulcer, and intramural hematoma-we have further explored refined classifications, including acute high-risk types and localized contrast enhancement of the aortic wall. For patients with different subtypes and at different stages of dissection-such as hyperacute, acute, or subacute-it is critical to develop individualized treatment strategies. These may include optimal medical therapy, isolated proximal endovascular repair, or combined proximal repair with distal bare stent implantation. Therefore, a large-scale clinical study is urgently needed to identify the optimal timing and approach for intervention based on refined classification schemes, and to establish personalized, stratified treatment strategies for different patient groups.

This project aims to conduct a real-world, prospective, multicenter, parallel-controlled study to compare outcomes between isolated proximal endovascular repair and combined proximal repair with distal bare stent implantation in patients with acute complicated or high-risk type B aortic dissection. The goal is to determine the most effective surgical approach for improving distal perfusion and promoting favorable aortic remodeling, thereby guiding treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged ≥18 years or non-pregnant female participants
* Diagnosed with acute complicated type B aortic dissection (defined as rupture/imminent rupture, associated ischemic syndromes [bowel, renal, or lower limb ischemia], radiologic progression of dissection or aortic dilation during hospitalization, uncontrolled hypertension, or refractory pain lasting over 12 hours), or high-risk type B dissection (defined as total aortic diameter >40 mm, false lumen diameter >22 mm, primary entry tear >10 mm, entry on the inner curvature, hemothorax, radiologic signs of ischemia [bowel, renal, or lower limb], or recurrent pain/symptoms).
* Patients deemed suitable for TEVAR or TEVAR combined with supra-aortic single-branch endovascular repair, as assessed by the investigator
* Patients who understand the purpose of the study, voluntarily agree to participate by signing informed consent, and are willing to comply with follow-up requirements

Exclusion Criteria:

* Subjects with hemodynamic instability or ruptured aortic dissection
* Subjects who, due to anatomical factors, are unsuitable for isolated TEVAR or TEVAR combined with supra-aortic single-branch reconstruction
* Subjects with connective tissue disorders, such as Marfan syndrome
* Subjects in poor general condition who cannot tolerate general anesthesia
* Subjects with known allergies to contrast agents or stent materials such as nitinol
* Subjects with a life expectancy of less than 12 months
* Subjects with a history of myocardial infarction or unstable angina within the past 3 months
* Subjects with a history of TIA or cerebral infarction within the past 3 months
* Subjects with serum creatinine levels >2.5 times the upper limit of normal or currently on dialysis
* Subjects with severe comorbidities such as liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population: Patients with type B aortic dissection receiving real-world clinical diagnosis and treatment at each participating center.
  Definition of Acute Complicated Type B Aortic Dissection:
  Patients diagnosed with type B aortic dissection within 14 days of symptom onset who present with rupture/imminent rupture, associated ischemic syndromes (bowel, renal, or lower limb ischemia), radiologic progression of dissection or aortic dilation during hospitalization, uncontrolled hypertension, or refractory pain lasting more than 12 hours.
  Definition of Acute High-Risk Type B Aortic Dissection:
  Patients diagnosed with type B aortic dissection within 14 days of symptom onset who exhibit one or more of the following: total aortic diameter >40 mm, false lumen diameter >22 mm, primary entry tear >10 mm, entry tear located on the inner curvature, hemothorax, radiologic signs of ischemia (bowel, renal, or lower limb), or recurrent pain/symptoms.
Sampling Method: Probability Sample
Enrollment: 438 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
30-day Postoperative Positive Remodeling Rate of the Descending Thoracic Aorta | 30 days
  (Number of subjects with positive remodeling of the descending thoracic aorta at the 30-day postoperative visit / Total number of subjects who completed the 30-day postoperative visit) × 100%
12-month Postoperative Degree of Positive Remodeling of the Descending Thoracic Aorta | 12 months
  Positive aortic remodeling is defined as meeting at least one of the following criteria:
  A reduction in the maximum diameter or volume of the false lumen, accompanied by either a decrease or an increase of less than 5 mm in the total aortic diameter or volume;
  An increase in the maximum diameter or volume of the true lumen, accompanied by either a decrease or an increase of less than 5 mm in the total aortic diameter or volume;
  A reduction in the maximum aortic diameter (along with changes in the diameters of both the true and false lumens).
  Formula for calculating the degree of positive remodeling of the descending thoracic aorta at 12 months postoperatively:
  (Maximum true lumen diameter of the descending thoracic aorta at 12 months post-op / Maximum total lumen diameter at 12 months post-op) - (Preoperative maximum true lumen diameter / Preoperative maximum total lumen diameter of the descending thoracic aorta)

SECONDARY OUTCOMES:
3-month Postoperative Positive Remodeling Rate of the Descending Thoracic Aorta | 3 months
Incidence of Distal Stent-Induced New Entry (d-SINE) During Follow-up Incidence of Distal Stent-Induced New Entry (d-SINE) During Follow-up Incidence of Distal Stent-Induced New Entry (d-SINE) During Follow-up | 5 years
Rate of Visceral Arterial Branch Lumen Loss During Follow-up | 5 years
Degree of Positive Remodeling of the Abdominal Aorta During Follow-up Degree of Positive Remodeling of the Abdominal Aorta During Follow-up Degree of Positive Remodeling of the Abdominal Aorta During Follow-up | 5 years
All-Cause Mortality Rate During Follow-up | 5 years
Aortic-related Mortality Rate During Follow-up | 5 years
Aortic-related Reintervention Rate During Follow-up | 5 years

IPD SHARING:
Plan to Share IPD: No